CLINICAL TRIAL: NCT04637126
Title: Cardiac Output Measurement in Critically Ill Patient in Sinus Rhythm: a Comparison Between Transpulmonary Thermodilution and Transthoracic Echocardiography
Brief Title: Cardiac Output Monitoring by Transpulmonary Thermodilution and Transthoracic Echocardiography in Critically Ill Patients
Acronym: TPTD-TTE-SR
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/19/0494; 2019-A03239-48 (Other: IDRCB)
Record Dates: First submitted 2020-11-06; First posted 2020-11-19 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: Sinus Rhythm
Keywords: Cardiac output monitoring; Transthoracic echocardiography; Transpulmonary thermodilution; Intensive care

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- mechanically ventilated and sedated patients with sinus rhythm: all mechanically ventilated and sedated patients with sinus rhythm hospitalized in our ICU and fitted with an hemodynamic monitoring by thermodilution technique due to hemodynamic failure
  Interventions: Other: Cardiac output measurement by transpulmonary thermodilution and transthoracic echocardiography

INTERVENTIONS:
Other: Cardiac output measurement by transpulmonary thermodilution and transthoracic echocardiography — Cardiac output is measured for all patients with transpulmonary thermodilution TPTD and transthoracic echocardiography TTE according to the recommendations

SUMMARY:
Cardiac output monitoring is a key component for the diagnosis and management of critically ill patients. The two less invasive methods commonly used in intensive care are transthoracic echocardiography and transpulmonary thermodilution. The objective of this study is to compare accuracy and trending ability of CO measurement by TPTD and TTE in critically ill patients with sinus rhythm.

DETAILED DESCRIPTION:
TTE is an easy noninvasive device now recommended as the first evaluation of the patient in circulatory failure but it present some limits due to poor echogenicity of patients, operator-dependent variability and cannot provide continuous hemodynamic data. TPTD is an invasive technique for CO monitoring recommended especially in shock not responsive to initial therapy.

Few studies have evaluated the level of agreement of each method (TTE and TPTD) with the reference method (pulmonary artery catheter) but they have never been compared between them with strong statistical analysis in particular trending ability.

It could be interesting to determine the level of concordance of these two methods of CO monitoring and trend ability by TPTD relative to TTE.

The investigators hypothesize that CO-TPTD are concordant with those performed by TTE.

Mechanically ventilated patients requiring hemodynamic assessment will be included. CO-TPTD will be measured via intermittent thermodilution. Blindly, a second investigator will use standard-view TTE to estimate CO-TTE as the product of stroke volume and the heart rate obtained during the measurement the blood flow velocity (using a Doppler technique) at the left ventricular outflow tract. A second measurement will be done with the two devices after a fluid challenge when patient requires it to compare trending ability.

ELIGIBILITY:
Inclusion Criteria:

* mechanically ventilated and sedated patients
* with sinus rhythm
* hospitalized in Intensive Care Unit
* fitted with an hemodynamic monitoring by thermodilution technique due to hemodynamic failure

Exclusion Criteria:

* age under 18
* arrhythmia
* severe aortic regurgitation or stenosis
* intracardiac shunt
* poor echogenicity
* tamponade
* major subject to a legal protection regim.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mechanically ventilated patients requiring hemodynamic assessment
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2020-03-06 (Actual); Primary Completion 2021-02-10 (Actual); Study Completion 2021-02-10 (Actual)

PRIMARY OUTCOMES:
bias between cardiac output measurement by TPTD and by TTE | Day 0
  bias between cardiac output measurement by transthoracic echocardiography and transpulmonary thermodilution

SECONDARY OUTCOMES:
percentage error between cardiac output measurement by transthoracic echocardiography and transpulmonary thermodilution | Day 0
  percentage error between cardiac output measurement by transthoracic echocardiography and transpulmonary thermodilution
percentage error between the value of Cardiac Output measured with TTE (transthoracic echocardiography) and the value of Cardiac Output measured withTPTD (transpulmonary thermodilution) after a fluid challenge. | 15 minutes after inclusion
  percentage error between the value of Cardiac Output measured with TTE and the value of Cardiac Output measured withTPTD after a fluid challenge.
The ability of TPTD (transpulmonary thermodilution) to track Cardiac Output as measured with TTE (transthoracic echocardiography) | 15 minutes after inclusion
  The ability of TPTD to track Cardiac Output as measured with TTE.

CONTACTS AND LOCATIONS:
Overall Officials: Antoine ROUGET, PH, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital of Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No